CLINICAL TRIAL: NCT05509348
Title: SMART Optimization of a Parenting Program for Active-duty Families
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00015375; CDMRP-PT150093 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2019-07-16; First posted 2022-08-22 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Parenting
Keywords: Parenting; Military Families; Prevention

STUDY DESIGN:
Intervention Model Description: Sequential multiple assignment randomization trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1: ADAPT Workshop (Experimental): 2 - day long in-person workshops (7 hours each day). Workshops are 2 weeks apart.
  Interventions: Behavioral: Phase 1: ADAPT Workshop
- Phase 1: ADAPT Online (Experimental): 3 weeks are given to complete 12 online modules using a secure website. Online modules include skill video, practice video, summary sheets, mindfulness audio and exercise video, printable handouts and motivation questionnaire.
  Interventions: Behavioral: Phase 1: ADAPT Online
- Phase 2: ADAPT Group (Experimental): 3 - 2 hour long in-person group sessions. Group sessions are consecutive weeks.
  Interventions: Behavioral: Phase 2: ADAPT Group
- Phase 2: ADAPT Individual (Experimental): 3 - 1 1/2 hour in-person individual sessions. Sessions are consecutive weeks.
  Interventions: Behavioral: Phase 2: ADAPT Individual

INTERVENTIONS:
Behavioral: Phase 1: ADAPT Workshop — 2 day workshop
  Arms: Phase 1: ADAPT Workshop
Behavioral: Phase 1: ADAPT Online — Online curriculum
  Arms: Phase 1: ADAPT Online
Behavioral: Phase 2: ADAPT Group — 3 in person group sessions
  Arms: Phase 2: ADAPT Group
Behavioral: Phase 2: ADAPT Individual — 3 sessions in person one on one
  Arms: Phase 2: ADAPT Individual

SUMMARY:
The overarching goal of the "SMART Optimization of a Parenting Program for Active-Duty Families" study is to advance the "development, adaptation, efficiency or optimization, and testing of a prevention intervention by using a sequential, multiple assignment, randomized trial/SMART to test multiple components of an empirically-supported parent training prevention intervention - After Deployment Adaptive Parenting Tools (ADAPT) for active-duty families negotiating multiple deployments and high deployment OPTEMPO (an army program that provides critical responses).

DETAILED DESCRIPTION:
Deployment (and particularly high deployment operational tempo/OPTEMPO) can generate family and personal stressors that disrupt supportive social relationships and functioning at home, thereby weakening the strength of military force in the field. Stressors include separation from, and reunification with families, concerns about mobilizations and combat stressors. These stressors, in turn, are associated with reduced parenting effectiveness, marital/partner difficulties, emotion dysregulation, and increased coercion. Coercion predicts risk for child maladjustment, as well as marital disruptions. Without effective prevention interventions, such environments may contribute to high divorce rates, child maladjustment, and reductions in service member wellbeing.

Most prevention interventions use a one-size-fits-all approach (i.e. all participants receive the same dose, format, and type of program) but this approach is often inefficient. Some families benefit from this approach but many do not. Adaptive interventions maximize efficiency, scalability, and sustainability, by providing families with a tailored dose, timing, program format, and/or sequence to improve outcomes based on their preferences and needs.

After Deployment: Adaptive Parenting Tools (ADAPT) is a Parent Management Training-Oregon (PMTO) program for military families with children ages 5-12 years old. PMTO is a theoretically-based family of interventions with extensive research supporting efficacy and effectiveness. ADAPT was developed and tested primary with National Guard/Reserve families. Program findings, based on 3 RCTs, indicate positive outcomes. No empirically supported parent training programs have been validated in RCTs for active duty military families with school-aged children in regular and high deployment OPTEMPO contexts.

The investigators are proposing a Phase III Clinical trial. The SMART optimization of a parenting program for active-duty families uses an adaptive intervention strategy to optimize an evidence-based universal prevention intervention, After Deployment Adaptive Parenting Tools/(ADAPT). SMART trials are rapidly gaining recognition within the medical and mental health fields as an innovative approach to developing adaptive treatment regimens. SMARTs have been successfully implemented in diverse areas including interventions for cancer, autism spectrum disorders, adolescent depression, and alcoholism. SMARTs also show considerable promise in innovating intervention approaches within prevention contexts.

In this study, the investigators will compress and test a variety of formats, sequences, and doses of ADAPT. The investigators will provide two 'first line' ADAPT programs and two slightly more intensive booster ADAPT programs for families who do not 'respond' to the first line intervention. Adaptive intervention strategies involve decision rules that specify how the type or intensity of an intervention should change depending on participants' response on a predetermined indicator of initial progress within an intervention. Within a SMART, a measure of initial response is used following delivery of an intervention in order to evaluate each families' need for further intervention programming. In this way, programming is tailored to meet the needs of individual families by providing additional services only to those families who are likely to benefit. This measure of initial response is referred to as a primary tailoring variable. In the proposed study, the primary tailoring variable is parental locus of control, a key variable shown in prior studies to predict change in observed parenting effectiveness, as well as change in other outcomes (PTSD symptoms, suicidality, and child adjustment).

The tested formats, sequences, and doses of ADAPT include:

1. Begin with ADAPT Online. Parents exhibiting initial response receive continued access to online resources. Parents exhibiting non-response are stepped-up to booster individual face-to-face ADAPT.
2. Begin with ADAPT Online. Parents exhibiting initial response receive continued access to online resources. Parents exhibiting non-response are stepped -up to booster group-based ADAPT.
3. Begin with ADAPT condensed group (with online support). Parents exhibiting initial response receive continued access to online resources. Parents exhibiting non-response are stepped to booster group-based ADAPT.
4. Begin with ADAPT condensed group (with online support). Parents exhibiting initial response continue access to online resources. Parents exhibiting non-response are stepped-up to booster group-based ADAPT.

This approach allows families who do not need intensive services to receive appropriately brief services. Those higher-need families receive more intensive services.

To address Aim 1, the investigators will compress the ADAPT group and individual curriculum, through consultation with service members, spouse, and content experts. The investigators will conduct two focus groups with parents who have returned from deployment (including spouses) and live on military installations and will assemble a Panel of 7 experts via a video conference call to inform program modifications. Each of the two parent focus group will consist of 12 families (24 individuals), one group at Fort Bragg with Special Operations (SO) participants, one group at Joint Base Lewis-McChord (JBLM) and Ft. Campbell with 12 Regular Army (RA) participants. To ensure gender sensitivity, the investigators will recruit and ask similar questions of mothers and fathers.

The investigators will ask an Expert Panel to view and advise on modifications to the current ADAPT NG/R group and individual materials. After reviewing the report of the focus group results, an Expert Panel will gather via videoconference (Month 4). Panel experts will weigh in on the results and be provided with two weeks to provide written recommendations. Expert panel and focus group feedback will inform (i) how to best compress key ADAPT skills, and (ii) address issues specific to high deployment OPTEMPO conditions. The focus group data and panel feedback will be used to finalize components for the SMART.

To address Aims 2,3,4: Among 210 SO and 315 RA families (i.e., total N=525 families) with 5-12 year-old children, the investigators will examine effects of ADAPT modalities and sequences/timing on multiple behaviors and outcomes (i.e., (i) coercive family interactions, positive parenting, couple adjustment, and co-parenting, (ii) parents PTSD symptoms, depression symptoms, substance use, (iii) child behavior and emotional problems, and positive adjustment, by conducting a 2-stage SMART, and (iv) document participation, satisfaction, and fidelity. To assess behaviors and outcomes, the investigators will administer and collect a series of assessments at 4 timepoints.

For Aims 2, 3, and 4, the investigators will use a 2-stage SMART design to examine the optimal sequence, dosage, and delivery formats of ADAPT for active duty military families living in a range of operational tempo contexts. The investigators will recruit a total of 525 families living on three installations: FT Bragg, FTs Belvoir/Myer and FT Campbell, with 210 families recruited from FTs Bragg and Campbell, and 105 from FTs Belvoir/Myer.

ELIGIBILITY:
Inclusion Criteria:

* families in which one parent has returned from deployment
* families with at least one child age 5 to 12 in their custody and living with parent(s) in the home
* must agree to randomization
* must indicate willingness to interact with study materials and complete assessment batteries

Exclusion Criteria:

* families with children younger than 5 or older than 12
* families in which at least one parent has an active psychosis
* families with an open child protection case for abuse or neglect in the family
* families in which there is a child with a serious mental health diagnosis (i.e., autism, child psychosis)
* youth who have a documented pervasive developmental disability or mental retardation
* families who participated in the focus group
* those with less than a 5th grade comprehension level in English

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Change in Observed Parenting Effectiveness | T1 (baseline), T3 (1 year) and T4 (2 years). Change is being assessed, primarily change between T1 and T3.
  Family Interaction Tasks (FIT) with each parent and child

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Gewirtz, PhD, Principal Investigator — University of Minnesota and Arizona State University
Locations (4):
- United States (4):
  - Fort Campbell, Fort Campbell North, Kentucky
  - Fort Bragg, Fort Bragg, North Carolina
  - Fort Myer, Arlington, Virginia
  - Fort Belvoir, Fort Belvoir, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almirall D, Compton SN, Gunlicks-Stoessel M, Duan N, Murphy SA. Designing a pilot sequential multiple assignment randomized trial for developing an adaptive treatment strategy. Stat Med. 2012 Jul 30;31(17):1887-902. doi: 10.1002/sim.4512. Epub 2012 Mar 22. PMID 22438190
- [Background] Kasari C, Kaiser A, Goods K, Nietfeld J, Mathy P, Landa R, Murphy S, Almirall D. Communication interventions for minimally verbal children with autism: a sequential multiple assignment randomized trial. J Am Acad Child Adolesc Psychiatry. 2014 Jun;53(6):635-46. doi: 10.1016/j.jaac.2014.01.019. Epub 2014 Mar 12. PMID 24839882
- [Background] Thall PF, Logothetis C, Pagliaro LC, Wen S, Brown MA, Williams D, Millikan RE. Adaptive therapy for androgen-independent prostate cancer: a randomized selection trial of four regimens. J Natl Cancer Inst. 2007 Nov 7;99(21):1613-22. doi: 10.1093/jnci/djm189. Epub 2007 Oct 30. PMID 17971530
- [Background] Murphy SA, Lynch KG, Oslin D, McKay JR, TenHave T. Developing adaptive treatment strategies in substance abuse research. Drug Alcohol Depend. 2007 May;88 Suppl 2(Suppl 2):S24-30. doi: 10.1016/j.drugalcdep.2006.09.008. Epub 2006 Oct 23. PMID 17056207
- [Background] August GJ, Piehler TF, Bloomquist ML. Being "SMART" About Adolescent Conduct Problems Prevention: Executing a SMART Pilot Study in a Juvenile Diversion Agency. J Clin Child Adolesc Psychol. 2016 Jul-Aug;45(4):495-509. doi: 10.1080/15374416.2014.945212. Epub 2014 Sep 25. PMID 25256135
- See also: ADAPT Program Website and Recruitment/Enrollment — http://adapt.umn.edu

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT05509348/Prot_SAP_000.pdf